CLINICAL TRIAL: NCT02735122
Title: A Randomized, Double-Blind, Placebo- and Active- Controlled, Single-Dose, Efficacy, Safety, and Pharmacokinetics Study of a Test Acetaminophen 500 mg Tablet in Postoperative Dental Pain
Brief Title: Study of Acetaminophen (ACM) in Post-operative Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Collaborators: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-151027203834-PACT
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Post Operative Dental Pain
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Test acetaminophen (Experimental): acetaminophen tablet and placebo caplet and placebo liquid-filled capsule
  Interventions: Drug: acetaminophen Tablet; Drug: Placebo Caplet; Drug: Placebo Liquid-filled capsule
- Commercial acetaminophen (Active Comparator): acetaminophen caplet and placebo tablet and placebo liquid-filled capsule
  Interventions: Drug: acetaminophen Caplet; Drug: Placebo Tablet; Drug: Placebo Liquid-filled capsule
- Commercial ibuprofen (Active Comparator): ibuprofen liquid-filled capsule and placebo tablet and placebo caplet
  Interventions: Drug: ibuprofen Liquid-filled capsule; Drug: Placebo Tablet; Drug: Placebo Caplet
- Placebo (Placebo Comparator): Placebo tablet and placebo caplet and placebo liquid-filled capsule
  Interventions: Drug: Placebo Tablet; Drug: Placebo Caplet; Drug: Placebo Liquid-filled capsule

INTERVENTIONS:
Drug: acetaminophen Tablet — 2 test acetaminophen 500 mg tablets
  Other Names: Test ACM
  Arms: Test acetaminophen
Drug: acetaminophen Caplet — 2 commercial acetaminophen 500 mg caplets
  Other Names: Commercial ACM
  Arms: Commercial acetaminophen
Drug: ibuprofen Liquid-filled capsule — 2 commercial ibuprofen 200 mg Liquid-filled capsules
  Other Names: Commercial IBU
  Arms: Commercial ibuprofen
Drug: Placebo Tablet — 2 placebo tablets
  Arms: Commercial acetaminophen; Commercial ibuprofen; Placebo
Drug: Placebo Caplet — 2 placebo caplets
  Arms: Commercial ibuprofen; Placebo; Test acetaminophen
Drug: Placebo Liquid-filled capsule — 2 placebo Liquid-filled capsules
  Arms: Commercial acetaminophen; Placebo; Test acetaminophen

SUMMARY:
This is a Dental Pain Study which will evaluate the analgesic onset, efficacy and safety of 1000 mg acetaminophen as two Test acetaminophen 500 mg tablets, compared with commercial products of acetaminophen 1000 mg administered as two 500 mg caplets, and ibuprofen (IBU) 400 mg following third molar (wisdom tooth) extraction.

DETAILED DESCRIPTION:
This is a single-dose, randomized, double-blind, triple-dummy, placebo- and active controlled, parallel-group study to evaluate the analgesic onset, efficacy, and safety profile of Test acetaminophen 1000 mg compared with two commercial products over a six-hour period after third-molar extractions. Subjects will undergo dental extraction of three or four third molars.

ELIGIBILITY:
Inclusion Criteria:

1. 17 years to 50 years old
2. Weight 100 lbs or greater with a body mass index (BMI) 18-30 inclusive
3. Dental extraction of three or four molars
4. Experience moderate to severe pain after extraction of third molars
5. Females of childbearing age must be willing to use acceptable method of birth control

Exclusion Criteria:

1. Currently pregnant or planning to be pregnant or nursing a baby
2. Known allergy to acetaminophen (ACM) or non-steroidal anti-inflammatory drugs (NSAIDS)
3. Inability to swallow whole large tablets or capsules
4. Have other conditions that the investigator feels may impact subject's safety and/or the integrity of the study

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 420 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Time to first confirmed perceptible pain relief | 6 hours
  Minutes until confirmed first perceptible pain relief are achieved. Stopwatch is started after the subject takes the study medication. The subject is instructed to stop the stopwatch when they first begin to feel any pain relief. The first perceptible pain relief is confirmed if the subject also stopped the second stopwatch indicating meaningful pain relief.

SECONDARY OUTCOMES:
Percentage of subjects with confirmed perceptible relief from 30 minutes to successively earlier minutes in one-minute increments (Test ACM versus placebo) | 30 minutes or less
Risk ratios of confirmed perceptible relief by 10 minutes (Test acetominophen and commercial ibuprofen) | 10 minutes or less
  The risk ratios and confidence intervals for incidence of confirmed perceptible relief of Test ACM divided by commercial IBU will be presented for 10 minutes
Risk ratios of confirmed perceptible relief by 15 minutes (Test acetominophen and commercial ibuprofen) | 15 minutes or less
  The risk ratios and confidence intervals for incidence of confirmed perceptible relief of Test ACM divided by commercial IBU will be presented for 15 minutes
Risk ratios of confirmed perceptible relief by 20 minutes (Test acetominophen and commercial ibuprofen) | 20 minutes or less
  The risk ratios and confidence intervals for incidence of confirmed perceptible relief of Test ACM divided by commercial IBU will be presented for 20 minutes
Percentage of subjects with meaningful relief by 30 minutes | 30 minutes or less
Time to meaningful pain relief | 6 hours
  Minutes until meaningful pain relief are achieved. Stopwatch is started after the subject takes the study medication. The subjects are instructed to stop the stopwatch when the relief from the starting pain is meaningful to them.

CONTACTS AND LOCATIONS:
Overall Officials: Derek D. Muse, M.D., Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
At this time we do plan to share IPD through the YODA site. The specific individual participant data sets have not yet been determined.

REFERENCES:
- [Derived] Myers A, Gelotte C, Zuckerman A, Zimmerman B, Shenoy A, Qi D, Cooper SA. Analgesic onset and efficacy of a fast-acting formulation of acetaminophen in a postoperative dental impaction pain model. Curr Med Res Opin. 2024 Feb;40(2):267-277. doi: 10.1080/03007995.2023.2294946. Epub 2024 Jan 24. PMID 38124555